CLINICAL TRIAL: NCT06262256
Title: Effects of High-intensity Interval Training on Myocardial Strain in Patients With Metabolic Syndrome
Brief Title: Effects of High-intensity Interval Training on Myocardial Strain in Metabolic Syndrome Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Castilla-La Mancha (Other)
Collaborators: Complejo Hospitalario de Toledo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HIIT-GLS-METS
Record Dates: First submitted 2024-01-19; First posted 2024-02-15 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: High-Intensity Interval Training; Metabolic Syndrome; Myocardial Dysfunction
MeSH Terms: conditions — Metabolic Syndrome | interventions — High-Intensity Interval Training

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial with control group
Who Masked: Outcomes Assessor
Masking Description: Echocardiography evaluators will be masked about participant allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Regular medical treatment for patients with metabolic syndrome.
- High-intensity interval training (Experimental): Regular medical treatment for patients with metabolic syndrome plus, 16 weeks of high-intensity interval training (3-times/week, 50 min/session conducted on stationary bike).
  Interventions: Behavioral: High-intensity interval training

INTERVENTIONS:
Behavioral: High-intensity interval training — supervised exercise conducted on stationary bikes after individualized intensity prescription.
  Arms: High-intensity interval training

SUMMARY:
the effects of high-intensity interval training on myocardial function will be studied in a group of patients under medical treatment for the components of metabolic syndrome.

DETAILED DESCRIPTION:
Objective: To analyze the effects of high-intensity interval training (HIIT) on myocardial function of metabolic syndrome patients.

Methods and design. Randomized clinical trial with a control group. Project was developed in association with the regional general hospital. Pre and post-intervention evaluation after 16 weeks of training for the HIIT group.

Subjects: Recruited using adverts published on public medical center boards. Up to 30 subjects per group (HIIT and CONTROL) will be recruited (at least 20% women) Measurements. Echocardiography: Global longitudinal strain (GLS), Mitral filling parameters, myocardial dimensions, and myocardial wall thickness.

Cardiorespiratory fitness: Maximal oxygen consumption, Maximal power output, Maximal oxygen pulse.

Clinical: Metabolic syndrome components and derived variables (e.g., triglycerides/high-density lipoprotein ratio) Body composition by anthropometric measurements and dual-energy X-ray absorptiometry.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of metabolic syndrome.
* Capacity to exercise on a stationary bike
* Inhabitant of the province of Toledo

Exclusion Criteria:

* Untreated cardiovascular disease with hemodynamic instability
* Untreated respiratory disease, symptomatic.
* Untreated metabolic disease.
* Untreated renal disease requiring dialysis.
* Contraindications for high-intensity exercise training

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2023-12-22 (Actual)

PRIMARY OUTCOMES:
Changes in global longitudinal strain | up to 16 weeks
  response to myocardial strain after intervention. Assessed by echocardiography, measured as a percentage

SECONDARY OUTCOMES:
changes in cardiorespiratory fitness | up to 16 weeks
  changes in maximal oxygen consumption measured in litres/min, all assessed by a cardiopulmonary exercise test in cycle-ergometer with breath by breath gas analysis.
changes in metabolic syndrome z-score | up to 16 weeks
  Adimensional variable used to assess in a unified score, the changes in the components of metabolic syndrome. The z-score is based on the cut-off points ot the components(fasting serum concentrations of glucose, triglycerides, and high density lipoprotein, all measured in mg/DL), waist circumference measured in cm, systolic and diastolic blood pressure measured in mm Hg), and the variance of each variable among participants assessed by the standard deviation.
changes in visceral fat | up to 16 weeks
  changes in visceral fat after intervention, assessed by dual-energy x-ray absortiometry. Measured in kg.
changes in left ventricle passive filling (E wave) | up to 16 weeks
  changes in early diastolic mitral inflow velocity (E wave), assessed by echocardiography. Measured in m/seg.
changes in early diastolic mitral annulus velocity (e' wave) | up to 16 weeks
  changes in early diastolic mitral annulus velocity (e' wave), assessed by echocardiography. Measured in m/seg.
changes in estimated left ventricle filling pressures (E/e') | up to 16 weeks
  changes in estimated left ventricle filling pressures by E/e' ratio (Peak E-wave velocity divided by the peak e' velocity) obtained by echocardiography, being E and e' measured in m/seg.

CONTACTS AND LOCATIONS:
Overall Officials: Juan F Ortega Fonseca, MD, Principal Investigator — University of Castilla-La Mancha
Locations (1):
- University of Castilla-La Mancha, Toledo, Castille-La Mancha, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] McDonagh TA, Metra M, Adamo M, Gardner RS, Baumbach A, Bohm M, Burri H, Butler J, Celutkiene J, Chioncel O, Cleland JGF, Coats AJS, Crespo-Leiro MG, Farmakis D, Gilard M, Heymans S, Hoes AW, Jaarsma T, Jankowska EA, Lainscak M, Lam CSP, Lyon AR, McMurray JJV, Mebazaa A, Mindham R, Muneretto C, Francesco Piepoli M, Price S, Rosano GMC, Ruschitzka F, Kathrine Skibelund A; ESC Scientific Document Group. 2021 ESC Guidelines for the diagnosis and treatment of acute and chronic heart failure. Eur Heart J. 2021 Sep 21;42(36):3599-3726. doi: 10.1093/eurheartj/ehab368. No abstract available. PMID 34447992
- [Result] Li C, Ford ES, McGuire LC, Mokdad AH. Association of metabolic syndrome and insulin resistance with congestive heart failure: findings from the Third National Health and Nutrition Examination Survey. J Epidemiol Community Health. 2007 Jan;61(1):67-73. doi: 10.1136/jech.2006.048173. PMID 17183018
- [Result] Crendal E, Walther G, Vinet A, Dutheil F, Naughton G, Lesourd B, Chapier R, Rupp T, Courteix D, Obert P. Myocardial deformation and twist mechanics in adults with metabolic syndrome: impact of cumulative metabolic burden. Obesity (Silver Spring). 2013 Dec;21(12):E679-86. doi: 10.1002/oby.20537. Epub 2013 Aug 23. PMID 23804526
- [Result] Mora-Rodriguez R, Ortega JF, Hamouti N, Fernandez-Elias VE, Canete Garcia-Prieto J, Guadalupe-Grau A, Saborido A, Martin-Garcia M, Guio de Prada V, Ara I, Martinez-Vizcaino V. Time-course effects of aerobic interval training and detraining in patients with metabolic syndrome. Nutr Metab Cardiovasc Dis. 2014 Jul;24(7):792-8. doi: 10.1016/j.numecd.2014.01.011. Epub 2014 Jan 29. PMID 24656853
- [Result] Smith BE, Peterman JE, Harber MP, Imboden MT, Fleenor BS, Kaminsky LA, Whaley MH. Change in Metabolic Syndrome and Cardiorespiratory Fitness Following Exercise Training - The Ball State Adult Fitness Longitudinal Lifestyle Study (BALL ST). Diabetes Metab Syndr Obes. 2022 May 20;15:1553-1562. doi: 10.2147/DMSO.S352490. eCollection 2022. PMID 35619799
- [Result] Murray J, Bennett H, Bezak E, Perry R, Boyle T. The effect of exercise on left ventricular global longitudinal strain. Eur J Appl Physiol. 2022 Jun;122(6):1397-1408. doi: 10.1007/s00421-022-04931-5. Epub 2022 Mar 16. PMID 35296909
- [Result] Serrano-Ferrer J, Crendal E, Walther G, Vinet A, Dutheil F, Naughton G, Lesourd B, Chapier R, Courteix D, Obert P. Effects of lifestyle intervention on left ventricular regional myocardial function in metabolic syndrome patients from the RESOLVE randomized trial. Metabolism. 2016 Sep;65(9):1350-60. doi: 10.1016/j.metabol.2016.05.006. Epub 2016 May 18. PMID 27506742
- [Result] Nagueh SF, Appleton CP, Gillebert TC, Marino PN, Oh JK, Smiseth OA, Waggoner AD, Flachskampf FA, Pellikka PA, Evangelisa A. Recommendations for the evaluation of left ventricular diastolic function by echocardiography. Eur J Echocardiogr. 2009 Mar;10(2):165-93. doi: 10.1093/ejechocard/jep007. No abstract available. PMID 19270053
- [Result] Asch FM, Miyoshi T, Addetia K, Citro R, Daimon M, Desale S, Fajardo PG, Kasliwal RR, Kirkpatrick JN, Monaghan MJ, Muraru D, Ogunyankin KO, Park SW, Ronderos RE, Sadeghpour A, Scalia GM, Takeuchi M, Tsang W, Tucay ES, Tude Rodrigues AC, Vivekanandan A, Zhang Y, Blitz A, Lang RM; WASE Investigators. Similarities and Differences in Left Ventricular Size and Function among Races and Nationalities: Results of the World Alliance Societies of Echocardiography Normal Values Study. J Am Soc Echocardiogr. 2019 Nov;32(11):1396-1406.e2. doi: 10.1016/j.echo.2019.08.012. PMID 31679581